CLINICAL TRIAL: NCT06480864
Title: Adebrelimab Plus Apatinib for Maintenance Treatment of Extensive Stage Small Cell Lung Cancer After First-line Induction with Adebrelimab Plus Chemotherapy (CLOG2402-ADAPT): a Multi-center, Single-arm, Phase 2 Clinical Trial
Brief Title: Adebrelimab Plus Apatinib for Maintenance Therapy of Extensive Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yunpeng Liu (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, Yunpeng Liu, Director, China Medical University, China
Organization: China Medical University, China (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-SCLC-LN-001
Record Dates: First submitted 2024-06-20; First posted 2024-06-28 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — apatinib; Carboplatin; Cisplatin; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adebrelimab+Chemotherapy→Adebrelimab+ Apatinib (Experimental): Participants will receive adebrelimab plus carboplatin /cisplatin and etoposide during the induction phase (4-6 cycles of three weeks.). Thereafter, participants will receive maintenance (after induction phase) adebrelimab plus apatinib until persistent PD, intolerable toxicity or withdrawal of consent.
  Interventions: Drug: Adebrelimab Injection; Drug: Apatinib Mesylate Tablets; Drug: Carboplatin; Drug: Cisplatin; Drug: Etoposide

INTERVENTIONS:
Drug: Adebrelimab Injection — Adebrelimab injection (1200mg) will be administered by intravenous infusion during the induction phase and maintenance phase on day 1 in a 3-week treatment cycle.
Drug: Apatinib Mesylate Tablets — Apatinib mesylate tablets (250 mg) will be administered orally in a 3-week treatment cycle, once a day.
Drug: Carboplatin — Carboplatin (AUC 4-5mg/mL/min) intravenous infusion will be administered during the induction phase on day 1 in a 3-week treatment cycle.
Drug: Cisplatin — Cisplatin (75mg/m2) intravenous infusion will be administered during the induction phase on day 1 in a 3-week treatment cycle.
Drug: Etoposide — Etoposide(100mg/m2) intravenous infusion will be administered during the induction phase from day 1 to 3 in a 3-week treatment cycle.

SUMMARY:
To evaluate the efficacy and safety of maintenance therapy with Adebrelimab plus Apatinib for extensive stage small cell lung cancer after first-line induction of Adebrelimab plus chemotherapy.

DETAILED DESCRIPTION:
This is a prospective, single-arm trial. To evaluate the efficacy and safety of maintenance therapy with Adebrelimab plus Apatinib for extensive stage small cell lung cancer after first-line induction of Adebrelimab plus chemotherapy.

Induction Period: Participants received adebrelimab (1200 mg, iv., Day1) + carboplatin (AUC 4-5 mg/mL/min)/cisplatin (75 mg/m2) + etoposide (100 mg/m2, D1-3) for 4-6 cycles of three weeks.

Maintenance phase: Participants received adebrelimab (1200mg, iv., Day1) + apatinib (250mg, po., daily) once every three weeks.

Follow-up: After disease progression, at the discretion of the investigator, apatinib and adebrelimab can be used across lines:

For platinum-sensitive patients (≥3 months from last chemotherapy): apatinib and adebrelimab plus platinum-containing two-agent chemotherapy (irinotecan/purple shirts in combination with platinum); for patients with PFS1 >12 months: chemotherapy can be continued with the original EC/EP regimen; For platinum-resistant patients (<3 months from last chemotherapy): apatinib and adebrelimab plus concurrent single-agent chemotherapy (irinotecan or single-agent purple shirts). The dose of chemotherapy agents was adjusted empirically by the investigators.

The primary endpoint is progression-free survival (PFS). Secondary endpoints include objective remission rate (ORR), disease control rate (DCR), duration of remission (DoR), and overall survival (OS); PFS2 (defined as time from enrolment to second disease progression or death) Our study will also explore biomarkers including: haematopoietic factors (IL-6,IL-8, IL-10, etc.), PD-L1 expression, T-cell subsets, T-cell immunoprecision typing and regulatory T-cell counts. The data from our study will provide the basis for further prospective clinical trials (Phase III).

ELIGIBILITY:
Inclusion Criteria:

1. Participants voluntarily enrolled in this study and signed an informed consent form, were compliant and co-operated with follow-up visits;
2. Age 18 years and above, male and female;
3. Diagnosis of extensive stage small cell lung cancer (ES-SCLC) confirmed by histology or pathology (according to the American Veterans Lung Cancer Association, VALG stage);
4. ECOG physical condition score is 0-2;
5. Subjects have not received systematic treatment for ES-SCLC in the past (including chemotherapy, VEGFR inhibitors and immune checkpoint inhibitors, etc.)
6. Patients with limited stage small cell lung cancer (LS-SCLC) who have received radiotherapy, chemotherapy or radiochemotherapy require a treatment-free period of more than 6 months. Patients with asymptomatic brain metastases are allowed to have cranial radiotherapy during induction chemotherapy;
7. Life expectancy >= 3 months;
8. There must be a measurable target lesion that meets the RECIST 1.1 criteria (CT scan length of the tumour lesion >10mm);
9. The function of major organs is normal, that is, the following criteria are met.

   * Blood routine (not transfused, not using haematopoietic factors and not corrected with drugs within 14 days): ANC ≥ 1.5 x 109/L; HB ≥ 90 g/L; PLT ≥ 100 × 109/L;
   * Biochemical tests:

   TBIL ≤ 1.5ULN; TBIL ≤ 1.5 ULN; ALT, AST ≤ 2.5 ULN;

   - Renal function: Serum creatinine (Cr) ≤ 1.5 x ULN or creatinine clearance ≥ 40 mL/min. (apply the standard Cockcroft-Gault formula):

   - Coagulation function must meet: INR ≤ 1.5 and APTT ≤ 1.5 ULN;
10. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to the first dose. Female subjects of childbearing potential and male subjects whose partner is a female of childbearing potential must agree to use a highly effective method of contraception and breastfeeding for the duration of the study up to 90 days after the last administration of study drug. The Investigator or his/her designee, in consultation with the subject, will be required to confirm that the subject has knowledge of how to properly and consistently use the contraceptive method;
11. For males, surgical sterilisation or agreement to use a highly effective method of contraception for the duration of the trial and for 90 days after the final administration of study drug;
12. For female participants, agreement to refrain from breastfeeding for the duration of the study or for 180 days after the last dose of study treatment is required.

Exclusion Criteria:

1. Patients with meningeal metastases;
2. Prior treatment with any T-cell co-stimulation or immune checkpoint therapy, including, but not limited to, cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) inhibitors, PD-1 inhibitors, PD-L1/2 inhibitors, CD137 agonists, or other agents that target T cells;
3. Prior treatment with apatinib;
4. Factors affecting oral administration of medications such as inability to swallow, post gastrointestinal resection, chronic diarrhoea, intestinal obstruction;
5. Any active autoimmune disease or history of autoimmune disease (e.g., uveitis, enteritis, hepatitis, pituitary gland inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (may be included after hormone replacement therapy), tuberculosis); and skin disorders (e.g., vitiligo, psoriasis, or alopecia) in which asthma has been in complete remission in childhood and has required no intervention in adulthood or in which systemic therapy is not required. or alopecia areata) may be included; patients requiring medical intervention with bronchodilators may not be included;
6. Patients with congenital or acquired immune function defects such as human immunodeficiency virus (HIV) infection, active hepatitis B (HBV DNA ≥ 500 IU/ml), hepatitis C (hepatitis C antibody positive with HCV-RNA above the lower limit of detection of the analytical method), or co-infection with both hepatitis B and hepatitis C;
7. Urine routine suggesting urinary protein ≥ (++), or 24h urine protein amount ≥ 1g or severe hepatic or renal insufficiency;
8. Subjects requiring systemic therapy with corticosteroids (>10 mg/day of prednisone or equivalent) or other immunosuppressive agents within 14 days prior to first dose. Inhaled or topical corticosteroids and adrenal hormone replacement therapy at doses > 10 mg/day prednisone efficacy dose are permitted in the absence of active autoimmune disease;
9. Subjects who have been treated with antitumour vaccines or other antitumour agents with immunostimulatory effects (interferon, interleukin, thymidine, immune cell therapy, etc.) within 1 month prior to the first dose;
10. Concomitant other malignancies ≤5 years prior to enrolment, except adequately treatable carcinoma in situ of the cervix, basal cell or squamous epithelial cell skin cancer, localised prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
11. Evidence of previous or current pulmonary fibrosis, interstitial pneumonitis, pneumoconiosis, radiographic pneumonia, drug-induced pneumonia, active pneumonia confirmed by imaging, and severely impaired lung function;
12. Uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg despite optimal pharmacological treatment);
13. Myocardial ischaemia or myocardial infarction of class II or greater, poorly controlled arrhythmias (including QTc intervals ≥450 ms in men and ≥470 ms in women). Myocardial infarction, New York Heart Association class II or higher heart failure, uncontrolled angina pectoris, uncontrolled severe ventricular arrhythmia, clinically significant pericardial disease, or electrocardiogram suggestive of acute ischaemia or active pericardial disease, within 6 months prior to enrolment, according to NYHA criteria, class III-IV cardiac insufficiency or cardiac ultrasound suggestive of a left ventricular ejection fraction (LVEF) of < 50% conduction system abnormalities;
14. Complicated severe infection within 4 weeks prior to first dose or unexplained fever >38.5°C during screening/prior to first dose;
15. Major surgery, open biopsy or significant trauma within 28 days prior to enrolment;
16. An arterial/venous thrombotic event within 6 months;
17. A significant risk of coughing up blood, bleeding events, or perforation as assessed by the investigator;
18. Known history of allogeneic organ transplantation or allogeneic haematopoietic stem cell transplantation;
19. Pregnant or lactating women; patients of childbearing potential who are unwilling or unable to use effective contraception;
20. Known hypersensitivity, hypersensitivity or intolerance to adebelizumab, apatinib, chemotherapeutic agents or their excipients;
21. Any condition which, in the opinion of the Investigator, may be detrimental to the subject or result in the subject's inability to meet or perform the requirements of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor by Resist1.1 (In months)

SECONDARY OUTCOMES:
Objective response rate (ORR) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor by Resist1.1 (In percent)
Disease control rate (DCR) | baseline up to approximately 6 month
  To evaluate the efficacy of anti-tumor by Resist1.1(In percent)
Duration of Response (DOR) | baseline up to approximately 12 months
  To evaluate the efficacy of anti-tumor by Resist1.1(In months)
Overall survival (OS) | baseline up to approximately 12 month
  To evaluate the efficacy of anti-tumor by Resist1.1(In months)
Second progression-free survival (PFS2) | baseline up to approximately 12 months
  To evaluate the efficacy of anti-tumor by Resist1.1(In months)
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From the initiation of the first dose to 28 days after the last dose
  To identify the incidence of AE and SAE in clinical trial

OTHER OUTCOMES:
Correlation of biomarkers and tumour response | baseline up to approximately 12 months
  Biomarkers Include: haematopoietic factors in pg/mL (IL-6,IL-8, IL-10, etc.), PD-L1 expression in TPS, T-cell subsets in percent, T-cell immunoprecision typing and regulatory T-cell counts in percent.

CONTACTS AND LOCATIONS:
Overall Officials: Xiujuan Qu, Principal Investigator — First Hospital of China Medical University
Locations (2):
- China (2):
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical University, Shenyang